CLINICAL TRIAL: NCT05513235
Title: Feasibility Study of a Mobile Digital Personal Health Record for Family-Centered Care Coordination for Children and Youth With Special Healthcare Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00109514; R21HS028699 (AHRQ)
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Children, Only; Children and Youth With Special Healthcare Needs
Keywords: Care coordination; Digital health; Mobile application; Primary care

STUDY DESIGN:
Intervention Model Description: Non-randomized single group feasibility study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Parents of eligible children and youth with special healthcare needs will use a digital personal record mobile application to coordinate care for six months.
  Interventions: Other: Digital personal health record

INTERVENTIONS:
Other: Digital personal health record — The digital personal health record is a mobile application ('app') entitled Caremap. The mobile app will be downloaded and accessible by parents/caregivers to help coordinate care.

SUMMARY:
A Fast Healthcare Interoperability Resources (FHIR)-enabled digital personal health record mobile app has the potential to enhance care coordination for families of children and youth with special healthcare needs (CYSHCN) and to inform improvements in family-centered care coordination that will be highly impactful for populations of patients with complex health needs across the age spectrum.

The purpose of this study is to evaluate the feasibility of a digital personal health record (PHR) mobile application integrated with electronic health records by FHIR data standards to enhance care coordination for families of CYSHCN. The study will enroll 40 families (adult parents/caregivers) of CYSHCN in pediatric primary care clinics to use the digital PHR mobile application as a tool for coordinating their child's care over a 6-month period. Using a single group, non-randomized study design and convergent mixed methods analyses, the study will: (a) determine the feasibility of FHIR-enabled integration of the mobile application with electronic health records for care coordination; (b) identify barriers and facilitators to implementation in real-world settings; and (c) examine associations between level of app adoption by families and family-reported outcome measures.

DETAILED DESCRIPTION:
Coordinating complex care across multiple providers and services can be stressful and isolating for families of children and youth with special healthcare needs (CYSHCN); thus, better care coordination solutions are needed. Digital personal health records (PHRs) that allow families to securely access, manage, and share their child's health data across multiple information and electronic health record (EHR) systems are promising solutions. Fast Healthcare Interoperability Resources (FHIR)-an application programming interface (API) standard that represents and exchanges health information-are central to digital PHRs being able to fulfill their promise. Despite their importance, FHIR technologies are not yet widely adopted. The researchers previously collaborated with Boston Children's Hospital on development of Caremap, a FHIR-enabled digital PHR mobile app that was co-designed with families and clinicians, to coordinate care for CYSHCN. Caremap has been positively reviewed by families in preliminary testing, and this followup research will implement and evaluate the Caremap mobile app in a real-world setting.

The specific aims of the study are as follows:

1. Evaluate the feasibility of a digital PHR mobile application with FHIR-enabled EHR integration to coordinate care for CYSHCN.
2. Identify barriers and facilitators of mobile app implementation via a mixed-methods evaluation.
3. Explore associations between mobile app adoption by families and family-reported outcomes.

The study will enroll 40 families (adult parents/caregivers) of CYSHCN in pediatric primary care clinics to use the digital PHR mobile application as a tool for coordinating their child's care over a 6-month period. Using a mixed-methods design, researchers will evaluate quantitative feasibility data and qualitative data from semi-structured interviews with families and providers and family stakeholder engagement panels to identify implementation barriers and facilitators. Using pre/post analyses of baseline and 6-month family-reported survey measures, they will explore associations between app adoption and family-reported outcomes.

If successful, the findings will support a future multisite, randomized trial to evaluate the effectiveness of enhanced care coordination with a digital PHR mobile app compared to usual care coordination. Due to similarities in needs between CYSHCN and adults with multiple chronic conditions, the study's findings will inform improvements in family-centered care coordination that will be highly impactful for complex populations across the age spectrum.

ELIGIBILITY:
Inclusion:

* Adult parent/legal guardian (age 18 or older) who is a primary caregiver for a CYSHCN aged 0-16 years
* Established care for their child/youth at a participating Duke Pediatrics Primary Care clinic: North Durham, South Durham,Brier Creek or Duke Med-Peds Primary Care sites (established = one or more completed visits in the past 12 months at the clinic)
* High level of complex medical needs that could benefit from additional care coordination support (determined by clinical provider at the participating clinic site)
* Primary care provider enrolled in the study as a provider participant/clinical provider site champion
* Active Duke MyChart (online EHR patient portal) account
* Full proxy access activated/enabled for parent to the child/youth's medical record in Epic
* Apple iOS device compatible with Caremap app requirements at time of consent

Exclusion Criteria:

* Non-English speaking
* Patients living in long-term, congregate settings - e.g., living in institutionalized settings such as long-term care facility, nursing/long-term rehab facilities
* Child is a ward of the state
* Lacks requisite technology to access and use mobile app (e.g., device/tablet/smartphone, home internet, active Epic MyChart account)
* Lack of decision-making capacity (parent/caregiver or adult patient, clinician-determined)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Technical feasibility (FHIR data transfer EHR to app) | Up to 6 months
  Quantitative measurement of technical feasibility assessed by success rate of FHIR-enabled EHR data transfer to app
Technical feasibility (FHIR data transfer app to provider dashboard) | Up to 6 months
  Quantitative measurement of technical feasibility processes assessed by success rate of FHIR-enabled transfer of family-reported health insights from app to EHR provider dashboard
Implementation (feasibility) | End of study (6 months)
  User-reported surveys of implementation outcomes assessed by the Feasibility of Intervention Measure (FIM), a 4-item scale that assesses whether a given method or condition can be successfully used in a specific setting. Responses to all survey items use a 5-point Likert scale from minimum 1 (completely disagree) to maximum 5 (completely agree). Higher scores are correlated with more positive responses.
Implementation (acceptability) | End of study (6 months)
  User-reported surveys of implementation outcomes assessed by the Acceptability of Intervention Measure (AIM), a 4-item scale that assesses whether a treatment or condition is satisfactory or agreeable to stakeholders. Responses to all survey items use a 5-point Likert scale from minimum 1 (completely disagree) to maximum 5 (completely agree). Higher scores are correlated with more positive responses.
Implementation (appropriateness) | End of study (6 months)
  User-reported surveys of implementation outcomes assessed by the Intervention Appropriateness Measure (IAM), a 4-item scale that assesses perceived compatibility or fit of a treatment or condition for a given setting or issue. Responses to all survey items use a 5-point Likert scale from minimum 1 (completely disagree) to maximum 5 (completely agree). Higher scores are correlated with more positive responses.
Change in parent/caregiver-reported degree of care integration, as measured by Pediatric Integrated Care Survey (PIC) | Baseline, 6 months
  Parent/caregiver report of experiences with care integration will be measured using the validated core 19-item PICS instrument. A composite score is calculated separately for each of the 5 survey constructs: access, communication, family impact, care goal creation, and team functioning.
Change in health-related quality of life (HR-QOL) | Baseline, 3 months, 6 months
  Parent/caregiver report of child's health-related QOL using the 9-item PROMIS Global 7+2 HR-QOL instrument, as well as a 2-item instrument assessing parent/caregiver perspectives on the impact of the child's conditions on their own and the parent/caregiver's usual activities and routines
Change in usability, as measured by the System Usability Scale (SUS) (provider) | Baseline, 6 months
  Provider report of experience and usability of the mobile app's provider dashboard using the 10-item SUS. This scale assesses participants' views of the usability of the app using a 5-point Likert scale from strongly agree to strongly disagree. Baseline version assesses their views on how usable they think the app will be, while the post version assesses their views on how usable the app actually was.
Net promoter score (NPS) (provider) | End of study (6 months)
  Provider-reported degree to which they would recommend the mobile app for use by others. NPS is a single item that measures the loyalty of customers to a company. NPS scores are measured with a single-question survey and reported with a number from the range -100 to +100, a higher score is desirable.

SECONDARY OUTCOMES:
Change in usability, as measured by the System Usability Scale (SUS) (parent/caregiver) | Baseline, 6 months
  Parent/caregiver report of experience and usability of the mobile app using the 10-item SUS. This scale assesses participants' views of the usability of the app using a 5-point Likert scale from strongly agree to strongly disagree. Baseline version assesses their views on how usable they think the app will be, while the post version assesses their views on how usable the app actually was.
Change in caregiver strain, as measured by the Caregiver Strain Questionnaire (Short Form 7; CGSQ-SF7) | Baseline, 3 months, 6 months
  Parent/caregiver report of degree of strain experienced as a result of their child's health with responses on a 5-point scale (1=not a problem at all; 5=very much a problem).
Change in confidence in avoiding hospitalization | Baseline, 3 months, 6 months
  Parent/caregiver-reported confidence in ability to avoid unplanned hospitalization in the next one month
Net promoter score (NPS) (parent/caregiver) | End of study (6 months)
  Parent/caregiver-reported degree to which they would recommend the mobile app for use by others. NPS is a single item that measures the loyalty of customers to a company. NPS scores are measured with a single-question survey and reported with a number from the range -100 to +100, a higher score is desirable.
Change in global health status | Weekly, up to 6 months
  Parent/caregiver report of their child's overall health status on a single item: 1 (poor) to 10 (excellent) numeric rating scale.
Adoption (family engagement) | Up to 6 months
  Quantitative measurement of family engagement with the app, assessed by weekly app log-ins by families.
Adoption (provider engagement) | Up to 6 months
  Quantitative measurement of provider engagement, assessed by count of views of EHR provider dashboard.
Adoption (app prescriptions) | Up to 6 months
  Quantitative measurement of prescription of the app to patients, assessed by count of times mobile app prescribed by provider for use.

CONTACTS AND LOCATIONS:
Overall Officials: David Y Ming, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ming DY, Wong W, Jones KA, Antonelli RC, Gujral N, Gonzales S, Rogers U, Ratliff W, Shah N, King HA. Feasibility of Implementation of a Mobile Digital Personal Health Record to Coordinate Care for Children and Youth With Special Health Care Needs in Primary Care: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2023 Sep 20;12:e46847. doi: 10.2196/46847. PMID 37728977

DOCUMENTS (1):
  • Informed Consent Form (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT05513235/ICF_000.pdf